CLINICAL TRIAL: NCT01935661
Title: A Case Control Study to Evaluate the Cognitive and Brain Function of β-thalassemia Patients in EMEK MEDICAL CENTER Compare to Healthy Controls.
Brief Title: A Case Control Study to Evaluate the Cognitive and Brain Function of β-thalassemia Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 111-12-EMC
Record Dates: First submitted 2013-08-07; First posted 2013-09-05 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Thalassemia; Brain Function (Measured by ERP Level)
Keywords: Blood transfusion; Hemosiderosis; ERP
MeSH Terms: conditions — Thalassemia; Hemosiderosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
β-thalassemia syndromes are a group of hereditary disorders characterized by a genetic deficiency in the synthesis of beta-globin chains.

In recent studies done in β-thalassemia major patients abnormal iron deposition was evident using MRI in brain structures, cortex, putamen, and caudate nucleus . In most of the cases the neurological involvement is subclinical. Cognitive functioning was evaluated in beta thalassemia major, compared with healthy controls, using a neuropsychological battery including tests of abstract reasoning, attention, executive functions, language, constructional/visuospatial skills, and memory. Patients with beta thalassemia major, in particular those showing signs of hemosiderosis, had significantly impaired function in all neuropsychological tests. There was no relationship between cognitive performances and signs of deferoxamine toxicity, deferoxamine dosage, and levels of hemoglobin and ferritin. Event-related potentials (ERPs) are one of the most informative and dynamic methods of monitoring the information stream in the living brain. ERPs are linked in time with a physical or mental event, and are typically extracted from the scalp-recorded electroencephalogram (EEG) by means of signal averaging.

ERPs have been used in the assessment of cognitive function in several disorders, including anemia and iron deficiency anemia. However, literature regarding cognitive function and ERP activity in thalassemia patients is extremely limited, especially in adults.

The purpose of this study is to evaluate the cognitive and brain function in a group of 60 thalassemia patients and compare the results to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia major and intermedia patients older than 6 years treated at Emek Medical Center Afula Israel.
* healthy controls matched for age and ethnicity.

Exclusion Criteria:

* patients suffering from acute diseases.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 60 Thalasssemia major and intermedia patients. 60 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain function assessment evaluated by Event-related potentials (ERPs of the information stream in the brain of Thalassemia patients. | one year

SECONDARY OUTCOMES:
correlation between brain function evaluated by ERP measurements and Hemosiderosis parameters like ferritin levels, Iron transferrin and Saturation. | one year

OTHER OUTCOMES:
correlation between pre and post transfusion status related to the Hemoglobin concentration and brain function measured by ERP. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit - Emek Medical Center
Locations (1):
- Haemek Medical Center, Afula, Israel